CLINICAL TRIAL: NCT01674036
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Ascending Single Oral Doses of Genz-682452 With a Pilot Investigation of Food Effect in Healthy Adult Male Subjects.
Brief Title: Safety, Tolerability and Pharmacokinetics of Genz-682452 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZFD00111/GZFD00211; TDU12766/FED12767 (Other: Sanofi Study Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — venglustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (GZFD00111/TDU12766): Genz-682452 (Experimental): Participants will receive a single oral dose of Genz-682452. Six ascending single doses and an optional seventh dose under fasted conditions will be used.
  Interventions: Drug: Genz-682452
- Part 1 (GZFD00111/TDU12766): Placebo (Placebo Comparator): Participants will receive a single oral dose of placebo.
  Interventions: Drug: Placebo
- Part 2 (GZFD00211/FED12767): Genz-682452 (Experimental): Participants will receive two single doses of Genz-682452 separated by a 7-day wash-out period, one dose given under fed (standardized high-fat breakfast) and one under fasted conditions. The dose will be based on the blind review of the safety/tolerability/pharmacokinetic data of single dose level cohorts in Part 1.
  Interventions: Drug: Genz-682452

INTERVENTIONS:
Drug: Genz-682452 — Capsules for oral administration.
  Arms: Part 1 (GZFD00111/TDU12766): Genz-682452; Part 2 (GZFD00211/FED12767): Genz-682452
Drug: Placebo — Placebo to Genz-682452
  Arms: Part 1 (GZFD00111/TDU12766): Placebo

SUMMARY:
The objectives of this study are to assess the tolerability, safety and pharmacokinetic parameters of Genz-682452 in healthy adult males, in two parts.

Part 1 (GZFD00111TDU12766): double-blind, randomized, placebo-controlled, sequential ascending single dose study;

Part 2 (GZFD00211FED12767): open-label, randomized, 2-sequence, 2-period, 2-treatment crossover study with a minimum wash-out period; to obtain preliminary information on the pharmacokinetics, tolerability and safety of Genz-682452 after single oral doses in fed and fasted conditions.

Subjects are not allowed to participate in more than 1 part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50.0 and 100.0 kg, inclusive, body mass index between 18.0 and 32.0 kg/m^2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting.
* Blood donation, greater than 100 mL, within 2 months before inclusion.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse.
* Unable to stop smoking cigarettes during the study.
* Excessive consumption of beverages containing xanthine bases.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events in Part 1 | Up to 4 weeks
Number of participants with adverse events in Part 2 | Up to 5 weeks

SECONDARY OUTCOMES:
Pharmacokinetics Plasma Parameters for Part 1 as measured by Cmax, tmax, AUC last, AUC, t1/2z, Vss/F, CL/F | Day 1 through Day 5
Pharmacokinetics Urine Parameters for Part 1 as measured by assessment of Genz-682452 urinary excretion, Ae0-t, fe0-t | Day 1 through Day 5
Pharmacokinetics Plasma Parameters for Part 2 as measured by Cmax, tmax, tlag, AUC last, AUC, t1/2z | Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Peterschmitt MJ, Crawford NPS, Gaemers SJM, Ji AJ, Sharma J, Pham TT. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Oral Venglustat in Healthy Volunteers. Clin Pharmacol Drug Dev. 2021 Jan;10(1):86-98. doi: 10.1002/cpdd.865. Epub 2020 Aug 26. PMID 32851809